CLINICAL TRIAL: NCT06848348
Title: A Randomized, Double-Blind, Placebo Controlled, Multicenter, Efficacy and Safety Study of Halneuron in the Treatment of Chemotherapy-Induced Neuropathic Pain
Brief Title: Efficacy and Safety Study of Halneuron in the Treatment of Chemotherapy-Induced Neuropathic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dogwood Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HAL-CINP-203
Record Dates: First submitted 2025-02-03; First posted 2025-02-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy Induced Neuropathic Pain
Keywords: Neuropathic Pain; Chemotherapy; Pain; Neuropathy; Cancer; CIPN; CINP
MeSH Terms: conditions — Neuralgia; Pain; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Halneuron (Experimental): Halneuron
  Interventions: Drug: Halneuron

INTERVENTIONS:
Drug: Halneuron — Halneuron for Subcutaneous Injection
  Arms: Halneuron
Drug: Placebo — Placebo for Subcutaneous Injection
  Arms: Placebo

SUMMARY:
A randomized study to determine safety and efficacy of single subcutaneous (SC) administration of HAL treatment in patients with CINP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years.
* Neuropathic pain has been present and is attributed to platinum and/or taxane chemotherapy.
* Patient has received a cancer chemotherapy regimen that included taxanes and/or platinum and has no active or discernible disease progression.

Exclusion Criteria:

* Current neuropathic pain with symptoms similar to CINP but attributed to causes other than platinum or taxane chemotherapy.
* Patients who have received HAL at any time prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To explore the efficacy of Halneuron in the treatment of patients with Chemotherapy-Induced Neuropathic Pain | From enrollment to end of study at 4 weeks
  Change from Baseline in the weekly average of daily 24-hour pain intensity scores analyzed by percentage of responders among patients treated with Halneuron compared to Placebo
To explore the Safety of Halneuron in the treatment of patients with Chemotherapy-Induced Neuropathic Pain | From enrollment to end of study at 4 weeks
  Incidence of serious adverse events (SAEs), adverse events (AEs) and Adverse Events of Special Interests (AESIs)

SECONDARY OUTCOMES:
Responder analyses for patient global impression of change (PGIC) | Enrollment to end of study at week 4
  Change from baseline for patient global impression of change (PGIC) items
Determine benefits of Halneuron treatment on non-pain outcomes including sleep quality, fatigue and mood | Enrollment to end of study at week 4
  Change from baseline to week 4 on the PROMIS fatigue
Determine benefits of Halneuron treatment on non-pain outcomes including sleep quality, fatigue and mood | Enrollment to end of study at week 4
  Change from baseline to week 4 on PROMIS Sleep instrument
Determine benefits of Halneuron treatment on non-pain outcomes including sleep quality, fatigue and mood | Enrollment to end of study at week 4
  Change from baseline to week 4 on the domains of the PROMIS-29

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Central Recruiting Site, Sheffield, Alabama
  - Central Recruiting Site, Glendale, Arizona
  - Central Recruiting Site, Fair Oaks, California
  - Central Recruiting Site, Fountain Valley, California
  - Central Recruiting Site, Los Angeles, California
  - Central Recruiting Site, Santa Rosa, California
  - Central Recruiting Site, Wheat Ridge, Colorado
  - Central Recruiting Site, Jacksonville, Florida
  - Central Recruiting Site, Lakeland, Florida
  - Central Recruiting Site, Orlando, Florida
  - Central Recruiting Site, Port Charlotte, Florida
  - Central Recruiting Site, Tampa, Florida
  - Central Recruiting Site, Atlanta, Georgia
  - Central Recruiting Site, Gurnee, Illinois
  - Central Recruiting Site, Farmington, Michigan
  - Central Recruiting Site, Fenton, Missouri
  - Central Recruiting Site, Kansas City, Missouri
  - Central Recruiting Site, Las Vegas, Nevada
  - Central Recruiting Site, Garden City, New York
  - Central Recruiting Site, Williamsville, New York
  - Central Recruiting Site, Winston-Salem, North Carolina
  - Central Recruiting Site, Salt Lake City, Utah
  - Central Recruiting Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR